CLINICAL TRIAL: NCT06956001
Title: A Phase III, Randomized, Multicentre, Open Label Study to Assess the Efficacy and Safety of Firmonertinib Versus Platinum Based Chemotherapy as First-line Treatment for Locally Advanced or Metastatic Non-small Cell Lung Cancer Patients With EGFR PACC Mutation or EGFR l861q Mutation
Brief Title: Firmonertinib Versus Platinum Based Chemotherapy as First-line Treatment for NSCLC With EGFR PACC or EGFR l861q Mutation
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Allist Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALSC013AST2818
Record Dates: First submitted 2025-04-09; First posted 2025-05-02 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-03

CONDITIONS: EGFR; NSCLC (Advanced Non-small Cell Lung Cancer)
Keywords: firmonertinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Injections; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Firmonertinib (Experimental): Oral administration, 240mg, QD。
  Interventions: Drug: Firmonertinib Mesilate Tablets
- chemotherapy (Active Comparator): Pemetrexed Disodium for Injection： 500mg/m2, intravenous infusion. Cisplatin for injection：75 mg/m2， intravenous infusion. Carboplatin Injection：administered according to the AUC of 5 mg/ml, intravenous infusion.
  Interventions: Drug: Pemetrexed Disodium for Injection; Drug: Cisplatin for injection; Drug: Carboplatin Injection

INTERVENTIONS:
Drug: Firmonertinib Mesilate Tablets — Usage and dosage: oral, 240mg, QD。 Medication duration: 21 days as a cycle, until intolerable toxicity, loss of clinical benefit, disease progression (confirmed by BICR), death or other anti-tumor treatment (whichever occurs first).
  Arms: Firmonertinib
Drug: Pemetrexed Disodium for Injection — Usage and dosage: 500mg/m2, intravenous infusion. Medication duration: 21 days as a cycle, D1 administration, until the occurrence of intolerable toxicity, loss of clinical benefit, disease progression (confirmed by BICR), death or other anti-tumor treatment (whichever occurs first).
  Arms: chemotherapy
Drug: Cisplatin for injection — Usage and dosage: 75 mg/m2, i.v. Medication duration: 21 days as a cycle, D1 administration, up to 4 cycles.
  Arms: chemotherapy
Drug: Carboplatin Injection — Usage and dosage: give the drug according to AUC 5 mg/ml, intravenous drip.
  Medication duration: 21 days as a cycle, D1 administration, up to 4 cycles.
  Arms: chemotherapy

SUMMARY:
This study is a randomized, open, multicenter phase III clinical study, which aims to evaluate the efficacy and safety of firmonertinib mesylate compared with platinum based chemotherapy for patients with locally advanced or metastatic NSCLC who have not been treated with systemic antitumor therapy and carry EGFR PaCC mutation or EGFR l861q mutation.

Eligible patients were stratified by EGFR mutation type and CNS metastasis at the time of enrollment. Approximately 300 patients would be randomly assigned 1:1 to receive either firmonertinib mesylate (240mg, orally on an empty stomach daily) or platinum containing dual agent chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form (ICF).
2. Age ≥18 years at the time of ICF signing.
3. At least one measurable lesion per RECIST v1.1, meeting the following:

   * No prior local therapy (e.g., radiotherapy)
   * Not used for biopsy during screening
4. Histologically/cytologically confirmed non-squamous NSCLC, classified as:

   * Locally advanced (Stage IIIB/IIIC, unsuitable for curative surgery and/or definitive chemoradiotherapy)
   * Metastatic (Stage IV) (Based on UICC/AJCC 8th edition TNM staging)
5. Agreement to provide:

   * Recent tumor tissue (from untreated lesions)
   * Blood samples
   * Central lab-confirmed EGFR PACC or L861Q mutation (If tumor tissue is unavailable due to inaccessible lesions, sponsor consultation is required.)
6. No prior systemic therapy for advanced/metastatic NSCLC.

   * Allowed if: Prior (neo)adjuvant/definitive chemoradiotherapy completed ≥12 months before recurrence/progression
7. ECOG performance status 0-1.
8. Life expectancy ≥12 weeks.
9. Adequate bone marrow/organ function within 14 days before treatment (no transfusion/G-CSF within 2 weeks prior).
10. Women of childbearing potential (WOCBP):

    * Abstinence or contraception use
    * No egg donation
11. Non-sterilized males:

    * Abstinence or contraception use
    * No sperm donation
12. CNS metastases allowed if protocol-specified criteria are met.

Exclusion Criteria:

1. Histologically/cytologically confirmed tumor with >10% neuroendocrine carcinoma, sarcomatoid carcinoma, or squamous cell components.
2. Known ALK-positive, ROS1-positive, RET fusion-positive, NTRK fusion-positive, BRAF V600E mutation, MET exon 14 skipping mutation, or other targetable alterations with approved therapies.
3. Prior treatments including:

   1. Systemic anti-tumor therapy for advanced/metastatic NSCLC (e.g., chemotherapy/targeted/immunotherapy). Neoadjuvant/adjuvant therapy exceptions per Inclusion Criterion #6.
   2. >30 Gy thoracic radiotherapy within 6 months or non-thoracic radiotherapy within 4 weeks prior to first dose (brain radiotherapy exceptions per Inclusion Criterion #12).
   3. Any prior EGFR-targeted therapy (including investigational EGFR-TKIs, mAbs, bispecific antibodies, etc.).
   4. Strong CYP3A4 inhibitors within 7 days or inducers within 21 days prior to first dose.
   5. Anticancer traditional Chinese medicines within 2 weeks prior to first dose.
   6. Non-specific immunomodulators (e.g., interferon, IL-2, thymosin) within 2 weeks prior to first dose.
   7. Major trauma/surgery within 4 weeks prior to treatment initiation.
4. Clinically significant gastrointestinal abnormalities, including:

   * Moderate/severe atrophic gastritis
   * GI obstruction/perforation
   * Chronic diarrhea/short bowel syndrome
   * Major upper GI surgery (e.g., gastrectomy)
   * Inflammatory bowel disease (Crohn's/ulcerative colitis) or active intestinal inflammation
   * Inability to swallow tablets
5. Uncontrolled systemic diseases.
6. Severe acute/chronic infections.
7. Interstitial lung disease (ILD)/non-infectious pneumonia:

   * History requiring clinical intervention
   * Current presence
   * Suspicious imaging findings unresolved at screening
8. Clinically significant cardiovascular dysfunction (active or history).
9. Tumor invasion of critical adjacent structures (heart/esophagus/SVC etc.) with high bleeding/fistula risk. Exceptions may be considered if investigator assesses minimal risk.
10. Pulmonary comorbidities causing severe impairment, including:

    1. Baseline lung diseases (e.g., pulmonary embolism [≤3 months], severe asthma/COPD/restrictive disease)
    2. Autoimmune/connective tissue disorders with pulmonary involvement (e.g., rheumatoid arthritis, sarcoidosis)
11. Residual toxicity >Grade 1 (per NCI CTCAE v5.0) from prior anticancer therapy (except alopecia/neuropathy).
12. Concurrent malignancies except:

    * Cured localized skin cancers (BCC/SCC), superficial bladder cancer, cervical/breast DCIS, or papillary thyroid cancer
    * Other malignancies cured by radical therapy ≥3 years prior
13. Pregnancy/lactation or planned pregnancy within 6 months post-treatment.
14. Inability to comply with study procedures/follow-up.
15. Known hypersensitivity to furmonertinib or excipients.
16. History of allergic reactions to pemetrexed/cisplatin/carboplatin.
17. Other exclusionary per investigator judgment, including:

    * Alcohol/drug abuse
    * Severe comorbidities (including psychiatric) requiring treatment
    * Critical laboratory abnormalities
    * Social/familial factors compromising safety/data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) assessed by the Independent Review Committee (BICR) according to RECIST v1.1. | Up to 3 years
  The time from the date of randomization to the date of first documentation of disease progression (assessed according to RECIST v1.1 criteria) or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 3 years
The incidence and severity of adverse events (AES) were determined according to NCI CTCAE V5.0 | Up to 3 years
Patient Reported Outcomes by EORTC QLQ LC13 questionnaire | Up to 3 years
  To assess the impact of firmonertinib on patients' disease-related symptoms and health related quality of life (HRQoL).
Patient Reported Outcomes by EORTC QLQ-C30 questionnaire | Up to 3 years
  To assess the impact of firmonertinib on patients' disease-related symptoms and health related quality of life (HRQoL).
Plasma concentrations of firmonertinib and its major metabolite (ast5902) in patients treated with firmonertinib at the indicated sampling time points | Up to 3 years

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Ethics Committee of cancer hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Shandong Tumor Hospital, Shandong, Jinan